CLINICAL TRIAL: NCT06772584
Title: Ginko Biloba Versus Desmopressin in Treatment of Children With Monosymptomatic Nocturnal Enuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Hossam Kandeel, Assistant lecturer of urology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5/2024UROL
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Enuresis, Nocturnal
Keywords: Nectornal enuresis
MeSH Terms: conditions — Nocturnal Enuresis | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Omegapress 0.2 (Active Comparator): Omegapress 0.2 was been taken by the pt
  Interventions: Drug: Desmopressin Acetate 0.2 mg Tablets
- Ginkobiloba (Active Comparator): Drug was taken by the pt
  Interventions: Drug: Ginkgobiloba
- Omegapress+ ginkgobiloba (Active Comparator): Both drugs were taken
  Interventions: Drug: Desmopressin Acetate 0.2 mg Tablets; Drug: Ginkgobiloba

INTERVENTIONS:
Drug: Desmopressin Acetate 0.2 mg Tablets — 3 groups of patients one received only desmopressin and group ginkobiloba ablnd group for both
  Arms: Omegapress 0.2; Omegapress+ ginkgobiloba
Drug: Ginkgobiloba — Group s take it as treatment of deep sleep in nectornal enuresis
  Arms: Ginkobiloba; Omegapress+ ginkgobiloba

SUMMARY:
Bedwetting among children is a common disorder, affecting 30% at age 4, 10% at age 6, 3% at age 12, and 1% at age.Untreated, the spontaneous cure rate is about 15% a year. Treatment is dominated by two approaches, enuresis alarm and drugs.

Treatment with drugs has largely been focused on tricyclic antidepressants especially imipramine or, more recently, antidiuretic agents such as desmopressin . For imipramine the proportion of total remission is 10-50% during treatment and a long term cure in 5-40%.8 However, numerous reports of side effects, some lethal, have led to a decline in its use.

Since Dimson in 1977 reported on the effects of desmopressinl" several double blind, placebo controlled studies have shown the efficacy of the drug often with rapid effect but also often with immediate relapse after ending treatment.

While one of theory of nocturnal enuresis is deep sleep in children , this the main cornerstone in using Alarm as line of management .

On the other hand drugs used in rehabitation of sleep rhythm seems to be with great benefits in management as GINKO BILOBA Ginkgo biloba leave extract is among the most widely sold herbal dietary supplements in the United States. Its purported biological effects include: scavenging free radical; lowering oxidative stress; reducing neural damages, reducing platelets aggregation; antiinflammation; anti-tumor activities; anti-aging , and improve night sleep rhythm

DETAILED DESCRIPTION:
Bedwetting among children is a common disorder, affecting 30% at age 4, 10% at age 6, 3% at age 12, and 1% at age.Untreated, the spontaneous cure rate is about 15% a year. Treatment is dominated by two approaches, enuresis alarm and drugs.

Treatment with drugs has largely been focused on tricyclic antidepressants especially imipramine or, more recently, antidiuretic agents such as desmopressin . For imipramine the proportion of total remission is 10-50% during treatment and a long term cure in 5-40%.8 However, numerous reports of side effects, some lethal, have led to a decline in its use.

Since Dimson in 1977 reported on the effects of desmopressinl" several double blind, placebo controlled studies have shown the efficacy of the drug often with rapid effect but also often with immediate relapse after ending treatment.

While one of theory of nocturnal enuresis is deep sleep in children , this the main cornerstone in using Alarm as line of management .

On the other hand drugs used in rehabitation of sleep rhythm seems to be with great benefits in management as GINKO BILOBA Ginkgo biloba leave extract is among the most widely sold herbal dietary supplements in the United States. Its purported biological effects include: scavenging free radical; lowering oxidative stress; reducing neural damages, reducing platelets aggregation; antiinflammation; anti-tumor activities; anti-aging , and improve night sleep rhythm

ELIGIBILITY:
Inclusion Criteria:

* All patients with monosymptomatic nocturnal enuresis

Exclusion Criteria:

* patients with day and night enuresis

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
To asses the effect of different drugs on number of bed time wetting | 3 months
  Drugs were administrated to the patient and response was documented regarding to number of bed wetting timed

CONTACTS AND LOCATIONS:
Locations (1):
- Menofia university, Cairo, State Or Province, Egypt